CLINICAL TRIAL: NCT06126471
Title: Prevalence and Pathological Features of C3 Dominant Glomerulonephritis Among Egyptian Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Ali Taha, Assistant lecturer of pathology, Sohag University
Other Study IDs: Soh-Med-23-10-12MD
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: C3 Nephropathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A classification has introduced C3 glomerulopathy (C3 glomerulopathy consensus report) that should be used to designate a disease process due to abnormal control of complement activation, deposition, or degradation and characterized by predominant glomerular C3 fragment deposits with EM dense deposits. Also, the consensus suggested that the term glomerulonephritis with dominant C3 should be used in practice as a morphological term for those cases with dominant C3 (C3c satining) which is defined as C3 intensity ≥ 2 orders of magnitude more than any other immune reactant on a scale of 0 to 3.

C3 glomerulonephritis with 3 dominant C3 deposits include C3 glomerulopathy, post-infectious glomerulonephritis (PIGN) and others such as para-protein associated glomerulonephritis.

In C3 glomerulopathy; the alternative pathway plays a major role in pathogenesis of this group of diseases. It occurs because of dysregulation of alternative complement pathway. Dysregulation can be due to mutations of complement proteins or to autoantibodies that promote complement activation.

Classical/lectin complement pathway has shown potential in evaluation of C3 glomerulopathy. It's suggested that presence of glomerular C4d which is a product of early classical/lectin pathway, should not exclude a C3 glomerulopathy.

Another disease group with prominent C3 deposits is postinfectious glomerulonephritis (PIGN) and although PIGN has traditionally been thought of as a disease triggered by glomerular immune complex deposition but C3 deposition in absence of immune complex deposits can be seen in patients with PIGN but with the emergence of C3 glomerulonephritis (C3GN), the distinction is difficult as the clinical and pathological presentation may be similar. However, their treatment and clinical course vary significantly.

In addition there is overlap between PIGN and C3 glomerulopathy as they may both show prominent sub-epithelial humps on electron microscopy. This overlap means that it may be very difficult to decide on morphology alone whether a biopsy is a typical PIGN that will resolve, or whether it represents a C3 glomerulopathy due to an underlying complement abnormality that will lead to persistent glomerulonephritis.

ELIGIBILITY:
Inclusion Criteria:

1. Adequate sample with at least 10 glomeruli
2. Enough residual tissues in the paraffin blocks
3. Available clinical data

Exclusion Criteria:

Other glomerular diseases such as lupus nephritis, IgA nephropathy, membranous glomerulonephritis and immune complex-mediated membranoproliferative GN. Cases of minimal change were also excluded.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Formalin-fixed and paraffin embedded renal tissue blocks from 100 patients.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To estimate the prevalence of C3 dominant glomerulonephritis | One or two days after staining sections with the markers
  C3 dominant glomerulonephritis

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Taha, Principal Investigator — Sohag university, faculty of medicine, Egypt
Locations (1):
- Sohag university , faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided